CLINICAL TRIAL: NCT06034041
Title: The Effect of Mediclore as an Anti-adhesion Agent and Safety in Full-endoscopic Spine Surgery: a Preliminary Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Nattapat Tangchitcharoen, Clinical Fellow in Spine Surgery, Chulalongkorn University, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 66
Record Dates: First submitted 2023-09-02; First posted 2023-09-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Disc Disease; Epidural Fibrosis; Failed Back Surgery Syndrome
MeSH Terms: conditions — Intervertebral disc disease; Failed Back Surgery Syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediclore (Experimental): After finish the operation, Mediclore group will be applied 1.5 CC of Mediclore at the surgical site. Mediclore is a Poloxamer-based thermosensitive anti-adhesive agent which is in a liquid solution and transform to a gel-state after being in a body temperature.
  Interventions: Drug: Mediclore
- Control (Placebo Comparator): After finish the operation, Control group will be applied 1.5 CC of normal saline at the surgical site.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Mediclore — After finish the operation, Mediclore group will be applied 1.5 CC of Mediclore at the surgical site. Mediclore is a Poloxamer-based thermosensitive anti-adhesive agent which is in a liquid solution and transform to a gel-state after being in a body temperature.
  Arms: Mediclore
Drug: Normal Saline — After finish the operation, Control group will be applied 1.5 CC of normal saline at the surgical site.
  Other Names: Control
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare efficacy and safety of Mediclore as anti-adhesion agent in patient who undergo endoscopic lumbar discectomy. The main question[s] it aims to answer are:

* efficacy (patient-reported outcomes, epidural fibrosis)
* safety (complications) Participants will received Mediclore at surgical site after finish the operation in experimental group and normal saline in control group.

Researchers will compare to see if experimental group have better patient-reported outcomes (PROs) after surgery with no different in complications rate.

DETAILED DESCRIPTION:
This study is a randomized clinical trial arrange in King Chulalongkorn Memorial Hospital. Participant will be randomly assigned into 2 groups by computer-generated sequence. Patients based-line characteristic data, patient-reported outcomes (VAS back/leg, ODI and EQ-5D) and a results of straight leg raising test will be collected. Participant will undergo a endoscopic lumbar discectomy by a singer spine surgeon. In experimental group, 1.5 CC. of Mediclore (poloxamer-based thermosensitive anti-adhesive agent) will be applied in after finish the operation. In control group normal saline 1.5 CC. will be applied instead.

Participants will proceed to regular follow-up protocol which include 1, 3 and 6 months visit at out-patient department. All of the PROs and a result of a straight leg raising test will be collected at each visit. MRI will be performed at 3 month after the surgery. The amount of epidural fibrosis will be evaluated according to Ross's method.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar disc herniated patients
* Failed proper conservative treatment more than 6 months

Exclusion Criteria:

* Previous history of lumbar spine surgery OR lumbar epidural steroid injection
* Infection OR malignancy
* Allergic to any given components
* Lactation and pregnency

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score for Leg pain (VAS Leg) | 3 month after surgery
  The VAS Leg consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('the worst pain in a lifetime'). The patient was asked to rate their current pain level by pointing the mark on the line.

SECONDARY OUTCOMES:
Visual Analogue Score for Leg and Back pain (VAS Leg, Back) | 1, 3 and 6 month after surgery (for VAS Back) and 1 and 6 month after surgery (for VAS Leg)
  The VAS Leg and Back consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('the worst pain in a lifetime'). The patient was asked to rate their current pain level by pointing the mark on the line.
Oswestry Disability Index (ODI) | 1, 3 and 6 month after surgery
  The ODI consists of 10 questions to assess the function in daily activities living, in which the responses are presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability).
EQ-5D-5L | 1, 3 and 6 month after surgery
  The EQ-5D-5L has 2 parts. In the first part, consist of 5 questions to assess the function in daily activities living, in which the responses are presented as 5 level (1 means no problems to 5 means extreme problems). The digits for the five questions can be combined into a 5-digit number that describes the patient's health state. The results will interpreted with the country specific utility score (Thailand) and reported as three decimal digit range from 0 (the worst health you can imagine) to 1 (the best health you can imagine).
Epidural Fibrosis | 3 month after surgery
  Evaluation of epidural fibrosis by method proposed by Ross et al (1999) by MRI. From MRI axial cut, A surgical intervertebral level will be marked as level 3, 2 adjacent cephalic image will be marked as level 1 and 2. 2 adjacent caudad level will be marked as level 4 and 5. Then each image will be separated into 4 quadrant. Fibrosis will be graded on a scale of 0-4 for each quadrant at each imaging slice encompassing the operative level: 0 = no/trace scar; 1 = > 0-25% of quadrant filled with scar; 2 = 25-50% of quadrant filled with scar; 3 = 50-75% of quadrant filled with scar; 4 = > 75% of quadrant filled with scar. The highest grade of epidural fibrosis from any image will represent the degree of epidural ficrosis.
Complication rate | peri-operation, 1, 3 and 6 month after surgery
Straight leg raising test | 1, 3 and 6 month after surgery
  Straight leg raising test will be performed at each visit. Results will be recorded as negative or positive. If positive, the degree that make a test positive will be also recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atlas SJ, Keller RB, Chang Y, Deyo RA, Singer DE. Surgical and nonsurgical management of sciatica secondary to a lumbar disc herniation: five-year outcomes from the Maine Lumbar Spine Study. Spine (Phila Pa 1976). 2001 May 15;26(10):1179-87. doi: 10.1097/00007632-200105150-00017. PMID 11413434
- [Background] Hansson E, Hansson T. The cost-utility of lumbar disc herniation surgery. Eur Spine J. 2007 Mar;16(3):329-37. doi: 10.1007/s00586-006-0131-y. Epub 2006 May 9. PMID 16683121
- [Background] Tosteson AN, Skinner JS, Tosteson TD, Lurie JD, Andersson GB, Berven S, Grove MR, Hanscom B, Blood EA, Weinstein JN. The cost effectiveness of surgical versus nonoperative treatment for lumbar disc herniation over two years: evidence from the Spine Patient Outcomes Research Trial (SPORT). Spine (Phila Pa 1976). 2008 Sep 1;33(19):2108-15. doi: 10.1097/brs.0b013e318182e390. PMID 18777603
- [Background] Loupasis GA, Stamos K, Katonis PG, Sapkas G, Korres DS, Hartofilakidis G. Seven- to 20-year outcome of lumbar discectomy. Spine (Phila Pa 1976). 1999 Nov 15;24(22):2313-7. doi: 10.1097/00007632-199911150-00005. PMID 10586454
- [Background] Asch HL, Lewis PJ, Moreland DB, Egnatchik JG, Yu YJ, Clabeaux DE, Hyland AH. Prospective multiple outcomes study of outpatient lumbar microdiscectomy: should 75 to 80% success rates be the norm? J Neurosurg. 2002 Jan;96(1 Suppl):34-44. doi: 10.3171/spi.2002.96.1.0034. PMID 11795712
- [Background] Ivanic GM, Pink TP, Homann NC, Scheitza W, Goyal S. The post-discectomy syndrome. Aetiology, diagnosis, treatment, prevention. Arch Orthop Trauma Surg. 2001 Oct;121(9):494-500. doi: 10.1007/s004020100289. PMID 11599749
- [Background] Hosseini S, Niakan A, Dehghankhalili M, Dehdab R, Shahjouei S, Rekabdar Y, Shaghaghian E, Shaghaghian A, Ghaffarpasand F. Effects of adhesion barrier gel on functional outcomes of patients with lumbar disc herniation surgery; A systematic review and meta-analysis of clinical trials. Heliyon. 2021 Jun 11;7(6):e07286. doi: 10.1016/j.heliyon.2021.e07286. eCollection 2021 Jun. PMID 34189319
- [Background] BenDebba M, Augustus van Alphen H, Long DM. Association between peridural scar and activity-related pain after lumbar discectomy. Neurol Res. 1999;21 Suppl 1:S37-42. doi: 10.1080/01616412.1999.11741025. PMID 10214570
- [Background] Ross JS, Robertson JT, Frederickson RC, Petrie JL, Obuchowski N, Modic MT, deTribolet N. Association between peridural scar and recurrent radicular pain after lumbar discectomy: magnetic resonance evaluation. ADCON-L European Study Group. Neurosurgery. 1996 Apr;38(4):855-61; discussion 861-3. PMID 8692415
- [Background] Ivanic GM, Pink PT, Schneider F, Stuecker M, Homann NC, Preidler KW. Prevention of epidural scarring after microdiscectomy: a randomized clinical trial comparing gel and expanded polytetrafluoroethylene membrane. Eur Spine J. 2006 Sep;15(9):1360-6. doi: 10.1007/s00586-006-0120-1. Epub 2006 Jun 9. PMID 16763848
- [Background] Guner D, Asik I, Ozgencil GE, Peker E, Erden MI. The Correlation of Epidural Fibrosis with Epiduroscopic and Radiologic Imaging for Chronic Pain after Back Surgery. Pain Physician. 2021 Dec;24(8):E1219-E1226. PMID 34793648
- [Background] Wang H, Sun W, Fu D, Shen Y, Chen YY, Wang LL. Update on biomaterials for prevention of epidural adhesion after lumbar laminectomy. J Orthop Translat. 2018 Mar 7;13:41-49. doi: 10.1016/j.jot.2018.02.001. eCollection 2018 Apr. PMID 29662790
- [Background] Gerszten PC, Moossy JJ, Flickinger JC, Welch WC. Low-dose radiotherapy for the inhibition of peridural fibrosis after reexploratory nerve root decompression for postlaminectomy syndrome. J Neurosurg. 2003 Oct;99(3 Suppl):271-7. doi: 10.3171/spi.2003.99.3.0271. PMID 14563144
- [Background] Du X, Wu L, Yan H, Jiang Z, Li S, Li W, Bai Y, Wang H, Cheng Z, Kong D, Wang L, Zhu M. Microchannelled alkylated chitosan sponge to treat noncompressible hemorrhages and facilitate wound healing. Nat Commun. 2021 Aug 5;12(1):4733. doi: 10.1038/s41467-021-24972-2. PMID 34354068
- [Background] Hajosch R, Suckfuell M, Oesser S, Ahlers M, Flechsenhar K, Schlosshauer B. A novel gelatin sponge for accelerated hemostasis. J Biomed Mater Res B Appl Biomater. 2010 Aug;94(2):372-379. doi: 10.1002/jbm.b.31663. PMID 20578223
- [Background] Zhao YF, Zhao JY, Hu WZ, Ma K, Chao Y, Sun PJ, Fu XB, Zhang H. Synthetic poly(vinyl alcohol)-chitosan as a new type of highly efficient hemostatic sponge with blood-triggered swelling and high biocompatibility. J Mater Chem B. 2019 Mar 21;7(11):1855-1866. doi: 10.1039/c8tb03181a. Epub 2019 Feb 21. PMID 32255048
- [Result] Ahn JH, Yoon SG, Yi JW, Kim SJ, Lee KE. Anti-adhesive effect and safety of a thermosensitive adhesion barrier (Mediclore) for thyroid surgery: a double-blinded randomized controlled trial. Ann Surg Treat Res. 2022 Jun;102(6):313-322. doi: 10.4174/astr.2022.102.6.313. Epub 2022 Jun 7. PMID 35800997
- [Result] Kim YI, Lee M, Kim SI, Seol A, Lee EJ, Kim HS, Song YS. A Randomized Controlled Trial of Thermo-Sensitive Sol-Gel Anti-Adhesion Agent after Gynecologic Surgery. J Clin Med. 2020 Jul 16;9(7):2261. doi: 10.3390/jcm9072261. PMID 32708699
- [Result] Chung JH, Kim KS, Choi JD, Kim TH, Lee KS, Oh CY, Noh JH, Kim JS, Kim WT, Lee SH, Kim JH, Kim TN, Huh W, Lee SW. Effects of poloxamer-based thermo-sensitive sol-gel agent on urethral stricture after transurethral resection of the prostate for benign prostatic hyperplasia: a multicentre, single-blinded, randomised controlled trial. BJU Int. 2020 Jan;125(1):160-167. doi: 10.1111/bju.14902. Epub 2019 Oct 6. PMID 31444917
- [Result] Choi HJ, Ryu JM, Chae BJ, Kim EK, Min JW, Shin HJ, Nam SJ, Yu J, Lee JE, Lee SK, Kim SW. Effect of Poloxamer-Based Thermo-Sensitive Sol-Gel Agent on Upper Limb Dysfunction after Axillary Lymph Node Dissection: A Double-Blind Randomized Clinical Trial. J Breast Cancer. 2021 Aug;24(4):367-376. doi: 10.4048/jbc.2021.24.e30. Epub 2021 Jun 17. PMID 34352935
- [Result] Shin SJ, Lee JH, So J, Min K. Anti-adhesive effect of poloxamer-based thermo-sensitive sol-gel in rabbit laminectomy model. J Mater Sci Mater Med. 2016 Nov;27(11):162. doi: 10.1007/s10856-016-5773-7. Epub 2016 Sep 19. PMID 27646404
- [Result] Fransen P. Reduction of postoperative pain after lumbar microdiscectomy with DuraSeal Xact Adhesion Barrier and Sealant System. Spine J. 2010 Sep;10(9):751-61. doi: 10.1016/j.spinee.2010.05.001. Epub 2010 Jun 12. PMID 20542472
- [Result] Ross JS, Obuchowski N, Modic MT. MR evaluation of epidural fibrosis: proposed grading system with intra- and inter-observer variability. Neurol Res. 1999;21 Suppl 1:S23-6. doi: 10.1080/01616412.1999.11758604. PMID 10214567